CLINICAL TRIAL: NCT01512641
Title: Prevalence of Dissociative Disorders in Children in a Population Supported in the Medico-social and Health Structures in Provence Alpes Cote d'Azur
Brief Title: Prevalence of Dissociative Disorders in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-API-01
Record Dates: First submitted 2011-12-13; First posted 2012-01-19 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Dissociative Disorders; Schizophrenia
Keywords: children dissociative disorders schizophrenia
MeSH Terms: conditions — Dissociative Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Children with Dissociative Disorders (Experimental): Children will take first the primary stage. If one child is positive, he will pass the secondary stage.
  Interventions: Other: Primary stage; Other: Secondary stage

INTERVENTIONS:
Other: Primary stage — Kiddie-Schedule for Affective Disorders and Schizophrenia
Other: Secondary stage — children who are positive to the kiddie-SADS (primary stage), will take the tests: PANSS, Scale for the Assessment of Negative Symptoms (SANS), ADI-R, scale TLC and WISC IV

SUMMARY:
Schizophrenia beginning before 18 years is a clinical entity not well known because of its low incidence and difficulties in the clinical diagnosis.

However, in the investigators clinical practice, due to the specialization of the investigators service, the investigators are led to hospital to receive important feel active of patients meeting the Diagnostic and Statistical Manual of Mental Disorders IV text revision (DSM IV-TR) precose schizophrenia.

The work of us team on the theme of the relationship between Pervasive Developmental Disorders and precose Schizophrenia led us to hypothesize that a number of children in care in the medical and educational institutes, hospitals and day shelters therapeutic part-time symptoms of schizophrenia or a line real early diagnosis of schizophrenia undervalued or not diagnosed.

The main goal is to estimate the prevalence of dissociative disorders in a population of children in care institutions and medical education in child psychiatry in hospitals and others structures.

ELIGIBILITY:
Inclusion Criteria:

* 7 to 18 years
* Supported in the partner institutions of the study
* IQ>35 on the certificate of orientation of the Maison Départementale des Personnes Handicapées (MDPH)
* Obtaining the agreement of parents and children

Exclusion Criteria:

* QI<35 on the certificate file Guidance MDPH
* Children not speaking french

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 301 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Rate of children diagnosed with dissociative disorders | between 2 and 4 hours depending children
  Rate of children diagnosed with dissociative disorders: children positive for the test Kiddie-Schedule for Affective Disorders and Schizophrenia (Kiddie-SADS).

SECONDARY OUTCOMES:
Percentage of children positive for test: Autism Diagnostic Interview-Revise (ADI-R). | 1 day on average
Scores of three dimensions of schizophrenia in the Positive And Negative Syndrome Scale (PANSS) | 4 hours
  3 dimensions: positive symptoms, negative symptoms and general psychopathology, based on these scores the diagnostic subtype of schizophrenia is established.
Score at the Test Lillois de Communication (TLC) | 30 minutes
Score on the Wechsler Intelligence Scale for Children-Fourth Edition (WISC IV)subtests and overall intelligence quotient (IQ). | 4 hours
Response time to test verbal fluency, scores on the Trail Making Test A (TMT) and TMT B. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Florence ASKENAZY, PU-PH, Study Director — University hospital of Nice; Emmanuelle DOR, PH, Principal Investigator — University hospital of Nice; François POINSO, PU-PH, Principal Investigator — AP-HM; Michèle BATTISTA, PH, Principal Investigator — Frejus's hospital; Michel BOUBLIL, PH, Principal Investigator — Antibes's hospital
Locations (4):
- France (4):
  - Psychiatrie infanto-juvénile - Centre Hospitalier d'Antibes, Antibes
  - Psychiatrie infanto-juvénile-Pôle femme-mère -enfant, Fréjus
  - Service de psychiatrie de l'enfant et de l'adolescent, Marseille
  - Service de psychiatrie de l'enfant et de l'adolescent, Nice

REFERENCES:
- [Derived] Dor-Nedonsel E, Menard ML, Fernandez A, Sakarovitch C, Fontas E, Salle-Collemiche X, Poinso F, Tosello AL, Maria F, Manera V, Askenazy F, Thummler S. Early-Onset Schizophrenia in a paediatric population of French psychiatric and medico-social care centres: A cross sectional study. PLoS One. 2020 Jul 27;15(7):e0236241. doi: 10.1371/journal.pone.0236241. eCollection 2020. PMID 32716957